CLINICAL TRIAL: NCT03701087
Title: Effect of Vitamin D Intake in Pregnancy to Prevent Recurrence of Gestational Diabetes
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, hadeer meshal, assistant professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: assistant professor
Record Dates: First submitted 2018-10-06; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Vitamin D Intake in First Trimester and Incidence of Gestational Diabetes Recurrence
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Effect of Vitamin D intake in pregnancy to prevent recurrence of gestational Diabetes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- normal serum vitamin D (No Intervention): normal serum vitamin D
- low serum level of vitamin D (Experimental): this arm will intake vitamin D 2800 IU daily
  Interventions: Drug: Vitamin D
- low serum vitamin D (Placebo Comparator): this arm will intake placebo omega 3
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — 2800 IU daily till 26 weeks of pregnancy
  Arms: low serum level of vitamin D; low serum vitamin D

SUMMARY:
primary outcome is vitamin D intake in first trimester for pregnant women with history of gestational diabetes in previous pregnancies and incidence of gestational diabetes recurrence secondary outcome is effect of vitamin D intake on mode of delivery, apgar score and neonatal birth weight

DETAILED DESCRIPTION:
it is a prospective randomized controlled study to determined the effect of vitamin D supplementation in pregnancy in reducing the incidence of gestational diabetes recurrence. it will be conducted at the department of obstetrics and gynecology kasr el ainy hospital faculty of medicine Cairo university from August 2018 to April 2020. we include in our study 430 pregnant women who had history of gestational diabetes in their previous pregnancies. patients with multiple pregnancy or with any medical disorder are excluded from study. BMI will be calculated for each participant at the time of admission and glucose challenge test will be performed for all patients in the first trimester to exclude diabetic patients from the study then a blood sample is taken from all patients enrolled in the study to measure the vitamin D level by ELISA (after fasting 12 hours and not have a fatty dinner) the participants will be assigned to one of three main groups according to the serum 25 OH vitamin D level. pregnant women with normal vitamin D level assigned as group A, pregnant women with lower serum level of vitamin D (>20 nmol/L) randomly divided into two groups: group B and C. Group B will be given oral vitamin D 2800 units daily till 26 week pregnancy and group C will be given Omega 3 as placebo till 26 week pregnancy. incidence of gestational diabetes will be measured in 24-26 week pregnancy with OGTT and compared in the three groups. All patients will be followed up till delivery. Mode of delivery, Apgar score and neonatal birth weight will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with history of gestational diabetes in previous pregnancies

Exclusion Criteria:

* multiple pregnancy
* pregnant patient with medical disorders

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 430 (Estimated)
Dates: Start 2018-08-02 (Actual); Primary Completion 2020-02-02 (Estimated); Study Completion 2020-04-02 (Estimated)

PRIMARY OUTCOMES:
incidence of gestational diabetes recurrence | 2 years
  incidence of gestational diabetes recurrence

CONTACTS AND LOCATIONS:
Overall Officials: ashraf mohsen, lecturer, Principal Investigator — Investigator
Locations (1):
- Kasr El Ainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No